CLINICAL TRIAL: NCT04419311
Title: Isokinetic Performance After Cruciate-substituting Ultra-congruent and Posterior Stabilized Total Knee Arthroplasties: A Randomized Controlled Trial
Brief Title: Isokinetic Performance After Cruciate-substituting Ultra-congruent and Posterior Stabilized Total Knee Arthroplasties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Erdem A Sezgin, Co-Principal Investigator, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1585/2017
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee; Knee Arthritis
Keywords: Ultra-congruent insert; Posterior cruciate ligament-stabilized insert; Isokinetic test; Strength; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients were randomized in a 1:1 ratio via computer-generated randomization using Microsoft Excel 2016 (Microsoft Corporation, Seattle, WA, USA) to be allocated in the UC insert or PS insert group before the TKA operation (Figure 1). Unblinded senior resident implemented the randomization. Patients and physiatrists performing isokinetic measurements were blinded to group allocation.
Who Masked: Participant, Investigator
Masking Description: Patients and physiatrists performing isokinetic measurements were blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ultra-congruent insert group (Experimental): Ultra-congruent inserts were used during total knee arthroplasty in patients randomized to this group.
  Interventions: Device: Vanguard® Knee System
- Posterior cruciate ligament-stabilized insert (Experimental): Posterior cruciate ligament-stabilized inserts were used during total knee arthroplasty in patients randomized to this group.
  Interventions: Device: Vanguard® Knee System

INTERVENTIONS:
Device: Vanguard® Knee System — Posterior cruciate ligament retention versus sacrificing is one of the main debates in total knee arthroplasty (TKA) and retention or sacrificing depends on the individual preference of the surgeon during the surgery. Whenever the surgeon decides to sacrifice the posterior cruciate ligament (PCL), another controversial question arises regarding the tibial insert type. While the posterior cruciate ligament-stabilized (PS) insert is widely used as the tibial insert in PCL-sacrificing TKA, it has some disadvantages such as increased polyethylene wear, additional bone resection, breakage of the post and patellar clunk syndrome. The ultra-congruent (UC) insert was designed to prevent bone loss in particular, and the other mentioned disadvantages of the conventional PS insert. However, patients with postoperative hyperextension have been seen to be associated with inferior clinical outcomes and knees become gradually more extended until two years after TKA using the UC insert.

SUMMARY:
The choice between ultra-congruent (UC) insert or posterior cruciate ligament-stabilized (PS) insert in posterior cruciate ligament (PCL) sacrificing total knee arthroplasty (TKA) remains debatable. Despite the potential advantages of the UC insert over PS insert with its different design, there are concerns about inferior clinical outcome related to its use. Therefore, isokinetic performance was used in this study to objectively evaluate knee function after TKA and the clinical scores of the patients were also evaluated. To the best of our knowledge, no prospective randomized study has compared the isokinetic performance of the knee following the use of UC and PS inserts in TKA. The hypothesis of the present study was that compared with the PS insert, the UC insert would be associated with a lower clinical outcome and isokinetic performance following TKA.

A total of 65 patients scheduled to undergo TKA on for primary knee osteoarthritis were randomly assigned to either the UC (32 patients) or the PS group (33 patients). The Knee Society Score (KSS) and isokinetic performance results of each patient were recorded preoperatively and at postoperative 3, 6 and 12 months. The physiatrist performing isokinetic tests and patients were blinded to the study.

DETAILED DESCRIPTION:
Eligibility of all patients between 55 and 80 years, scheduled to undergo unilateral TKA on for primary knee osteoarthritis will be evaluated. The exclusion criteria are rheumatological joint diseases, previous knee surgery, neuromuscular diseases, bilateral TKA, or insufficiency of collateral ligaments. Patients will be randomized in a 1:1 ratio via computer-generated randomization using Microsoft Excel 2016 (Microsoft Corporation, Seattle, WA, USA) to be allocated in the UC insert or PS insert group before the operation. Unblinded senior resident will implement the randomization. Patients and physiatrists performing isokinetic measurements will be blinded to group allocation.

During the UC and PS operations, Vanguard® Complete Knee System prosthesis (Zimmer Biomet Inc., Warsaw, IN, USA) will be implanted using the same surgical technique in all patients. The Vanguard anterior-stabilized (AS) insert is a UC deep-dish design with a 10 mm prominent anterior lip and 5mm posterior lip. This bone-conserving design prevents anterior femoral subluxation because of the prominent anterior lip. The insert design allows it to be used with the Vanguard cruciate-retaining femoral component and the highly congruent articulating surface increases rotational stability. There is more contact area between the femoral component and the weight-bearing surface to decrease the shear stress between the femur and polyethylene insert.

A tourniquet will be inflated to pressure of 300 mmHg after spinal anesthesia. All operations will be performed with the same surgical technique by a single senior surgeon. Patellar surface arthroplasty will be performed in all the cases. Both femoral and tibial prostheses will be implanted with pressured bone cement. A suction drain will be placed inside the knee capsule. On the morning of the first day after surgery patients will be mobilized under the supervision of the physical therapist. All patients will undergo the same rehabilitation procedure during the outpatient period and will be examined by the same physiatrist at the regular 3, 6, and 12-month follow-up visits.

The primary outcome is isokinetic performance, measured as peak knee extensor and flexor torque values in Newton-meters, on the operated knee. Measurements wilil be done preoperatively and at 3, 6, and 12-month follow-up examinations under the supervision of the same physiatrist. At same time points, the Knee Society Score (KSS) will be evaluated as well. Isokinetic measurements will be performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc., Shirley, NY, USA) by the same senior physiatrist. Patients will be positioned on the dynamometer with the hip in 90° in a sitting position for the knee flexion and extension measurements. Lateral movement of the knee will be prevented during full extension and flexion of the knee by a thigh strap on the operated leg. The physical therapist will help the patients to achieve proper positioning before each test. Concentric isokinetic knee flexion-extensions will be assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions will be completed by each patient. Instructions will be provided, and one trial repetition will then performed by all patients before the measurements were taken.

Sample size estimation will be performed using the extension peak torque as a primary effect variable. As there is no similar study with isokinetic measurements regarding this subject, a difference in mean values of 10 Nm and standard deviation of 12 Nm were assumed for each group. The group sample sizes of 31 and 31 achieved a power of 0.90 to detect a difference of 10 Nm between the two groups with estimated group standard deviations of 12 for each group and with a significance level (alpha) of 0.05 using a two-sided, two-sample test. Considering the loss to follow-up, two patients were added to each group. Thus, recruitment will end after 33 patients were assigned to either groups. All data will be calculated as mean and standard deviation. The Student's t-test will be used for statistical analysis of the patient data. Statistical calculations will be performed with SPSS 22.0 software (IBM SPSS Statistics for Windows, Version 22.0. Armonk, NY: IBM Corp.). A value of p< 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 80 years
* Scheduled to undergo unilateral TKA on for primary knee osteoarthritis

Exclusion Criteria:

* Rheumatological joint diseases
* Previous knee surgery
* Neuromuscular diseases
* Bilateral TKA
* Insufficiency of collateral ligaments

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Çankaya, MD, Principal Investigator — Aksaray University Training and Research Hospital
Locations (1):
- Aksaray University Training and Research Hospital, Aksaray, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Started | 33 | 33
Completed | 32 | 33
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.18 (8.55) | 67.67 (8.12) | 68.42 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 4 | 7 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Baseline Assessment of Peak Knee Extensor Torque Preoperatively
Description: Peak extensor torque values of each patient was recorded for the operated knee preoperatively under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
Newton meters | 55.56 (8.65) | 58.33 (8.96)

2. Primary Outcome: Baseline Assessment of Peak Knee Flexor Torque Preoperatively
Description: Peak flexor torque values of each patient was recorded for the operated knee preoperatively under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
Newton meters | 37.84 (9.56) | 40.3 (7.79)

3. Primary Outcome: Assessment of Peak Knee Extensor Torque at 3 Months Postoperatively
Description: Peak extensor torque values of each patient was recorded for the operated knee at postoperative 3 months under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
Newton meters | 44.38 (7.37) | 45.85 (7.46)

4. Primary Outcome: Assessment of Peak Knee Flexor Torque at 3 Months Postoperatively
Description: Peak flexor torque values of each patient was recorded for the operated knee at postoperative 3 months under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
Newton meters | 31.91 (10.11) | 29.39 (7.16)

5. Primary Outcome: Assessment of Peak Knee Extensor Torque at 6 Months Postoperatively
Description: Peak extensor torque values of each patient was recorded for the operated knee at postoperative 6 months under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).
Time Frame: 6 months postoperative
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
Newton meters | 53.53 (7.95) | 52.64 (6.83)

6. Primary Outcome: Assessment of Peak Knee Flexor Torque at 6 Months Postoperatively
Description: Peak flexor torque values of each patient was recorded for the operated knee at postoperative 6 months under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).
Time Frame: 6 months postoperative
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
Newton meters | 36.19 (9.86) | 35.27 (7.35)

7. Primary Outcome: Assessment of Peak Knee Extensor Torque at 12 Months Postoperatively
Description: Peak extensor torque values of each patient was recorded for the operated knee at postoperative 12 months under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).
Time Frame: 12 months postoperative
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
Newton meters | 59.34 (8.97) | 61.52 (9.88)

8. Primary Outcome: Assessment of Peak Knee Flexor Torque at 12 Months Postoperatively
Description: Peak flexor torque values of each patient was recorded for the operated knee at postoperative 12 months under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).
Time Frame: 12 months postoperative
Measure: Mean (Standard Deviation); unit: Newton meters
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
Newton meters | 39.94 (9.96) | 41.18 (7.63)

9. Secondary Outcome: Baseline Knee Society Clinical Score Evaluation
Description: The Knee Society Score were applied preoperatively.
  The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. The KSS Scale ranges from 0 to 200. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The KSCS ranges from 0 to 100. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. The KSFS ranges from 0 to 100. For each section, a score of 80-100 was considered excellent; 70-79, good; 60-69, fair; < 60, poor.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
score on a scale | 47.69 (12.6) | 49.15 (11.68)

10. Secondary Outcome: Knee Society Clinical Score Evaluation at 3 Months Postoperatively
Description: The Knee Society Clinical Score were applied at postoperative 3 months.
  The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. The KSS Scale ranges from 0 to 200. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The KSCS ranges from 0 to 100. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. The KSFS ranges from 0 to 100. For each section, a score of 80-100 was considered excellent; 70-79, good; 60-69, fair; < 60, poor.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
score on a scale | 78.81 (11.73) | 79.48 (10.80)

11. Secondary Outcome: Knee Society Clinical Score Evaluation at 6 Months Postoperatively
Description: The Knee Society Clinical Score were applied at postoperative 6 months.
  The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. The KSS Scale ranges from 0 to 200. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The KSCS ranges from 0 to 100. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. The KSFS ranges from 0 to 100. For each section, a score of 80-100 was considered excellent; 70-79, good; 60-69, fair; < 60, poor.
Time Frame: 6 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
score on a scale | 86.81 (5.64) | 88.39 (6.29)

12. Secondary Outcome: Knee Society Clinical Score Evaluation at 12 Months Postoperatively
Description: The Knee Society Clinical Score were applied at postoperative 12 months.
  The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. The KSS Scale ranges from 0 to 200. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The KSCS ranges from 0 to 100. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. The KSFS ranges from 0 to 100. For each section, a score of 80-100 was considered excellent; 70-79, good; 60-69, fair; < 60, poor.
Time Frame: 12 months postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
score on a scale | 90.69 (4.41) | 92.24 (4.44)

13. Secondary Outcome: Baseline Knee Society Functional Score Evaluation
Description: The Knee Society Functional Score were applied preoperatively.
  The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. The KSS Scale ranges from 0 to 200. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The KSCS ranges from 0 to 100. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. The KSFS ranges from 0 to 100. For each section, a score of 80-100 was considered excellent; 70-79, good; 60-69, fair; < 60, poor.
Time Frame: Preoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
units on a scale | 49.53 (14.11) | 51.27 (11.60)

14. Secondary Outcome: Knee Society Functional Score Evaluation at 3 Months Postoperatively
Description: The Knee Society Functional Score were applied at postoperative 3 months.
  The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. The KSS Scale ranges from 0 to 200. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The KSCS ranges from 0 to 100. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. The KSFS ranges from 0 to 100. For each section, a score of 80-100 was considered excellent; 70-79, good; 60-69, fair; < 60, poor.
Time Frame: 3 months postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
units on a scale | 64.47 (14.19) | 65.73 (11.90)

15. Secondary Outcome: Knee Society Functional Score Evaluation at 6 Months Postoperatively
Description: The Knee Society Functional Score were applied at postoperative 6 months.
  The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. The KSS Scale ranges from 0 to 200. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The KSCS ranges from 0 to 100. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. The KSFS ranges from 0 to 100. For each section, a score of 80-100 was considered excellent; 70-79, good; 60-69, fair; < 60, poor.
Time Frame: 6 months postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
units on a scale | 70.22 (12.98) | 72.21 (11.73)

16. Secondary Outcome: Knee Society Functional Score Evaluation at 12 Months Postoperatively
Description: The Knee Society Functional Score were applied at postoperative 12 months.
  The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. The KSS Scale ranges from 0 to 200. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The KSCS ranges from 0 to 100. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. The KSFS ranges from 0 to 100. For each section, a score of 80-100 was considered excellent; 70-79, good; 60-69, fair; < 60, poor.
Time Frame: 12 months postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
Number analyzed (Participants) | 32 | 33
units on a scale | 81.47 (10.45) | 82.79 (10.06)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Definition of adverse event does not differ from the clinicaltrials.gov definitions.
Arm/Group | Ultra-congruent Insert Group | Posterior Cruciate Ligament-stabilized Insert
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/32 | 2/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultra-congruent Insert Group (N=32) | Posterior Cruciate Ligament-stabilized Insert (N=33)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Superficial infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT04419311/Prot_SAP_001.pdf